CLINICAL TRIAL: NCT04271826
Title: Grey Zone Appendicitis (Intermediate Risk Alvarado Score 5-6): Role of Blood Test Biomarkers to Detect Early Appendicitis and to Decrease the Incidence of Negative Appendectomy: Cost and Effectiveness: Randomized Controlled Trial
Brief Title: Grey Zone Appendicitis: Role of Blood Test Biomarkers to Detect Early Appendicitis and to Decrease the Incidence of Negative Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zagu
Record Dates: First submitted 2020-02-09; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases with normal CT (Experimental): evaluate level of bilirubin and phospholipase A2 and their relation to positive or negative appendicitis
  Interventions: Procedure: laparoscopic appendectomy
- cases with proven appendicitis on CT (Experimental): evaluate level of bilirubin and phospholipase A2 and their relation to positive or negative appendicitis
  Interventions: Procedure: laparoscopic appendectomy

INTERVENTIONS:
Procedure: laparoscopic appendectomy — cases with normal CT underwent laparoscopic appendectomy

SUMMARY:
Introduction: many investigations emerged in the last decades and contribute towards a diagnosis of unsure appendicitis; they are valuable to the emergency general surgeon.

Aim: This study aims to assess the role of laboratory markers (bilirubin and phospholipase A2) individually or combined with Computed Tomography (CT) for the diagnosis of grey zone appendicitis (Alvarado score 5-6).

Methods: This prospective study included all 310 patients admitted with right iliac fossa (RIF) pain who had Alvarado score 5-6 (intermediate risk of appendicitis). All underwent full laboratory investigations including serum total bilirubin and phospholipase A2. All are underwent CT scan and classified into group A with normal CT but with persistent right iliac fossa pain and group B with proved acute appendicitis by CT. All cases underwent a laparoscopic or open appendectomy. Other causes of hyperbilirubine¬mia are excluded among the patients.

DETAILED DESCRIPTION:
INTRODUCTION Acute appendicitis is a very common surgical emergency worldwide, with a lifetime risk reported to be 7-8%..Accordingly, appendectomy is the most frequently performed operation worldwide.

Many surgical centers attempt to reduce surgical procedures performed during the night, and delaying appendectomy for 12-24 h does not seem to increase complications

Despite thorough research, the diagnosis of acute appendicitis is still difficult and remains the most common problem in clinical surgery.

In addition to clinical examination of the patients with appendicitis, ultrasonography and multidetector computed tomography (MDCT) have become the most useful tools with a respective sensitivity and specificity of 98.5% and 98.0% in expert centers Routine use of MDCT not only increases exposure to radiation but also very expensive and time-consuming. Thus evolving methods to diagnose early acute appendicitis without radiological examinations are of interest.

Observing serum bilirubin and phospholipase A2 level came into consideration as it seems to elevate in early appendicitis, its determination is fast and can be performed with other commonly performed blood tests.

Bacteria invade the appendix and release tumour necrosis factor-alpha, Interleukien 6, and cytokines. These substances reach the liver through superior mesenteric vein and cause dysfunction of liver either by direct effect or indirectly through altering the hepatic blood flow. So it is important to evaluate the total bilirubin level in the diagnosis of clinically suspected cases of appendicitis (6) THE AIM OF THE WORK

This study aims to evaluate the role of bilirubin and phospholipase A2 in:

1. Cases of grey zone unsure appendicitis (intermediate risk Alvarado score 5-6).
2. As a complementary to CT.
3. Detect early cases of appendicitis.
4. Decrease the incidence of negative appendicitis.
5. Decrease complications of missed cases of appendicitis.
6. Reduce the overnight appendectomy rate with its complications. Patients and methods Cases with normal CT but with persistent right iliac fossa tenderness and failed to improve under conservative treatment for 48 hrs With antibiotic therapy (Group A) underwent laparoscopic appendectomy. Patients proved to be appendicitis by CT underwent laparoscopic exploration (Group B). All the appendices removed were sent for histological examination and the operated cases divided into positive appendicitis (macroscopic or microscopic) and negative appendicitis.

Group A , patients with normal CT but with persistent right iliac fossa pain. Group B , patients with proved acute appendicitis in CT.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than 14years of both sexes.
* Non pregnant female.
* Patients taking analgesics. .Patients who diagnosed to have grey zone diagnosis of acute appendicitis (Alvarado score 5-6).

Exclusion Criteria:

* Alvarado score >6 or < 5.
* Cases of sure acute appendicitis.
* Documented Liver disease, biliary disease (congenital or acquired), hemolytic diseases and history of alcoholism.

  4) Cases revealed other pathology than appendicitis by CT and laparoscopy.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
serum bilirubin level | 1 year
  role of blood biomarker in detecting acute appendicitis
phospholipase A2 level | 1 year
  role of blood biomarker in detecting acute appendicitis

CONTACTS AND LOCATIONS:
Overall Officials: tamer A. alnaimy, MD, Principal Investigator — Zagazig University
Locations (1):
- Tamer Alsaied Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No